CLINICAL TRIAL: NCT00661050
Title: Exercise and Meditation: A Pilot Study of Alternative Techniques in the Treatment of Chronic Pelvic Pain Related to Painful Bladder Syndrome (PBS)/Interstitial Cystitis (IC) PI: Dr. Christopher Payne
Brief Title: Treatment of Interstitial Cystitis/Painful Bladder Syndrome Using Alternative Techniques: Exercise, Meditation, Tai Chi
Status: Withdrawn | Type: Observational
Why Stopped: Terminated due to low enrollment.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-03132008-1041; 11838
Record Dates: First submitted 2008-04-04; First posted 2008-04-18 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2011-03

CONDITIONS: Cystitis, Interstitial
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Alternative Medicine
Procedure: Tai Chi instruction and class participation or walking exercise and sitting meditation

SUMMARY:
Complementary and alternative medicine (CAM) is the term for medical products and/or practices that are not part of the current standard of care. Standard care is what medical doctors, doctors of osteopathy and allied health professionals, such as registered nurses and physical therapists, practice. Alternative medicine means treatments that you use instead of standard ones. Complementary medicine means nonstandard treatments that you use along with standard ones. The purpose of this study is to determine whether there is any improvement in symptoms reported by patients with chronic painful bladder syndrome when participating in alternative medical therapy/ exercise and meditative techniques. The specific alternative techniques participants will be randomized to in this trial include: Tai Chi instruction or walking exercise combined with sitting meditation.

DETAILED DESCRIPTION:
Participants will be referred for trial screening if they have a diagnosis of painful bladder syndrome/IC in the opinion of the investigator. Participants will be required to read the informed consent form and sign it prior to the screening of any medical information. The eligibility criteria will be reviewed and participants who qualify will complete the visit one study screening procedures. Participants will be asked to track there daily pain level and medication use for 7 days prior to randomization an in addition will be required to complete one 24-hour void diary during this same screening time period. Participants will be asked to give a urine sample on the day of screening and the day of randomization to screen for bladder infection. Female participants will be asked to provide a urine sample for pregnancy testing prior to randomization.

Participants will be required to be on a stable medical regime for 30 days prior to randomization. No new IC therapy or new pain treatments will be allowed to begin during the screening period and/or the 3 month study trial period. Participants will be allowed to continue on any IC/pain therapy they have used prior to screening.

Randomization to the treatment groups will occur 5-7 days prior to treatment start date. At that visit the patient#s medical history will be reviewed for eligibility and adverse events. The recorded pain scores collected and all quality of life measurements obtained. Participants who continue to qualify will be randomized to the specified treatment group.

Once 12 participants have been screened and are ready for randomization the participants will be scheduled for the randomization visit--Participants assigned to the Tai Chi group will be instructed on the logistics of the class, participants in this group will attend two classes/week- each class will be 1.5 hours in duration. The first 30 minutes will consist of standing meditation and progressive relaxation, the remaining 60 minutes will be TaiChi form instruction. The classes will meet bi-weekly for 3 months.

Participants will be contacted by the blinded coordinator at 2 week intervals to assess pain level, medication use, and adverse event monitoring, all data will be documented.

The exercise/meditation group will receive guided imagery CD and a pedometer to record the distance walked/bimonthly assessment. Participants will be asked to reserve 90 minutes twice weekly to complete the 30 min of walking exercise followed immediately by the 60 min of relaxation/mediation using the CD provided to them by the study. Participants will be asked to complete the exercise on the same days and times each week. The study coordinator will contact the participants every 2 weeks to assess pain level, medication use, and monitor for adverse events.

Participants will not be responsible for the costs of the Tai Chi classes, pedometer, and relaxation-guided imagery CD. Participants will be required to provide the CD player; patients will not be eligible if they do not have access to one. Participants will not be reimbursed for travel costs to the Tai Chi classes. Participants will be seen in clinic for the end-point evaluation 3-7 days after 3 month treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has signed and dated the appropriate Informed Consent document.
2. Participant is equal or > 18 years old
3. Participant has a clinical diagnosis of IC/PBS and or CP/CPPS in the opinion of the investigator
4. Participant with IC/PBS has reported a bladder pain or discomfort symptom score of 3 or greater on a 0-10 Likert scale over the previous four weeks. This bladder pain/discomfort criterion must be met at each of the two baseline screening visits as reported by the participant.
5. Participant with IC/PBS has reported a symptom score of abnormal urinary frequency of 3 or greater on 0-10 Likert scale over the previous four weeks. This frequency criterion must be met at least each of the two baseline screening visits.
6. Participant has had symptoms of discomfort or pain in the pelvic region for at least a three (3) month period within the last six (6) months.
7. Participant has previously undergone at least one course of other form of standard therapy for his/her symptoms Exclusion Criteria:1. Participant can not stand in place for at least 15 minutes.

Exclusion Criteria:

1. Participants have severe lower extremity disease that would prohibit participation in walking or Tai Chi movements.
2. Participant cannot hold urine for at least 30 minutes
3. Participant has relevant neurologic disorder that affects bladder and/or neuromuscular function in the opinion of the investigator.
4. Participant has active urethral or ureteral calculi, urethral diverticulum.
5. Participant has a history of pelvic radiation therapy, tuberculous cystitis, bladder cancer, carcinoma in situ, prostate cancer, or urethral cancer.
6. Participant has/reports any severe debilitating or urgent concurrent medical condition.
7. Participant has a potentially significant pelvic pathology or abnormalities on examination or prior imaging, including prolapse beyond the hymenal ring, pelvic mass, etc. that could cause or contribute to the clinical symptoms or require treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IC Patients from Stanford University Urology Clinic's patient population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Payne, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States